CLINICAL TRIAL: NCT07251803
Title: An Observational Study to Examine Non-inferiority of the Standard ASA Fasting Guidelines Versus 24-hour Clear Liquid Diet for Gastric Volume in Patients Taking GLP-1 Agonists
Brief Title: GLP1 Fasting Status and Gastric Retention Using Gastric Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Christopher Wolla, Assistant Professor-Faculty, Medical University of South Carolina
Other Study IDs: Pro00147318
Record Dates: First submitted 2025-11-11; First posted 2025-11-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Gastric Retention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASA fasting guidelines: Scheduled elective surgery and meet ASA fasting guidelines (NPO for at least 8 hours prior)
  Interventions: Diagnostic Test: Gastric Ultrasound
- 24-hour clear liquid diet: Scheduled elective colonoscopy and have been on a clear liquid diet for at least 24 hours prior
  Interventions: Diagnostic Test: Gastric Ultrasound

INTERVENTIONS:
Diagnostic Test: Gastric Ultrasound — All participants will undergo a gastric ultrasound in the preoperative area prior to their scheduled procedure. The patient will be placed in supine position. A curvilinear ultrasound probe will be placed on the sagittal plane below the xiphoid process. The probe will then slide along the costal margin to the right until the gastric antrum is identified. At this point, the ultrasound image will be obtained, and appropriate measurements will be taken. The patient will be placed in the right lateral decubitus position (RLD), and the above procedure will be repeated. The measurement of gastric antral cross-sectional area while in the RLD position will be recorded and used to calculate the gastric volume.

SUMMARY:
This study will enroll patients 18 years and older who are taking a GLP-1/GIP medication and 1) are scheduled for elective surgery and meet ASA fasting guidelines (nothing by mouth for at least 8 hours prior), or 2) scheduled elective colonoscopy and have been on a clear liquid diet for at least 24 hours prior. Participants will have a gastric ultrasound prior to surgery to measure any retained gastric contents. The purpose of this study is to determine if people taking GLP-1 receptor agonists and who fast normally are at an equal risk for having retained gastric contents after appropriately fasting for surgery, compared to patients who are on a liquid only diet for 24 hours prior to surgery.

DETAILED DESCRIPTION:
Patients will be classified into one of two groups:

1. Taking a GLP-1/GLP-GIP medication and undergoing an elective colonoscopy and have been on a clear liquid diet for the past 24-hours.

   or
2. Taking a GLP-1/GLP-GIP medication and undergoing am elective surgery and have fasted appropriately according to ASA guidelines.

All participants will undergo a gastric ultrasound in the preoperative area prior to their scheduled procedure. This will be completed to determine the amount of retained gastric contents, if any, after fasting properly prior to the procedure. An anesthesiologist attending who is properly trained on performing gastric ultrasounds and listed as a study team member will be the one performing the scan.

The patient will be placed in supine position. A curvilinear ultrasound probe will be placed on the sagittal plane below the xiphoid process. The probe will then slide along the costal margin to the right until the gastric antrum is identified. At this point, the ultrasound image will be obtained, and appropriate measurements will be taken. The patient will be placed in the right lateral decubitus position (RLD), and the above procedure will be repeated. The measurement of gastric antral cross-sectional area while in the RLD position will be recorded and used to calculate the gastric volume.

If based on the formula: GV (mL) = 27.0+(14.6*CSA)-(1.28*age) the patient is shown to have a gastric volume greater than 1.5mL/kg, or Antral Grade 2, the anesthesiologist assigned to the case will be alerted and will determine whether or not it is safe to continue with the scheduled surgery as the risk for aspiration may be higher based on the gastric ultrasound results.

Qualitative grading of the appearance of the gastric antrum in RLD will be graded as follows:

* Grade 0 antrum appears empty in both positions, and suggests no gastric content is present.
* Grade 1 antrum appears empty in the supine position, but clear fluid is visible in the RLD, consistent with a small volume of gastric fluid.
* Grade 2 antrum is that in which clear fluid is evident in both patient positions, or any solids in any position which is consistent with a higher volume state.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Have taken a GLP-1 or GLP-GIP agonist medication within the past 30 days
* ASA Physical Classification Status 1-3
* Fall into one of the following groups:

  1. Scheduled elective surgery and meet ASA fasting guidelines (NPO for at least 8 hours prior)
  2. Scheduled elective colonoscopy and have been on a clear liquid diet for at least 24 hours prior

Exclusion Criteria:

* Previous gastric or esophageal surgery
* Abnormal gastric anatomy
* Pregnancy
* Unable to provide written, informed consent
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will consist of patients who have taken a GLP-1 or GLP-GIP agonist medication within the past 30 days, and are scheduled for either an elective surgery and appropriately NPO for at least 8 hours prior, or scheduled for elective colonoscopy and have been on a clear liquid diet for at least 24 hours prior.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pre-operative gastric volume per unit of weight (ml/kg) as assessed by gastric ultrasound. | From enrollment until completion of pre-operative gastric ultrasound (typically within 3 hours of scheduled procedure).
  While the patient is in supine position, the gastric volume will be measured via ultrasound and then calculated using a validated formula, GV (mL) = 27.0+(14.6*CSA)-(1.28*age).

SECONDARY OUTCOMES:
Perlas antral grade | From enrollment until completion of gastric ultrasound (within 3 hours of scheduled procedure).
  Qualitative grading of the appearance of the gastric antrum in right lateral decubitus (RLD) will be graded as follows:1
  * Grade 0 antrum appears empty in both positions, and suggests no gastric content is present.
  * Grade 1 antrum appears empty in the supine position, but clear fluid is visible in the RLD, consistent with a small volume of gastric fluid.
  * Grade 2 antrum is that in which clear fluid is evident in both patient positions, or any solids in any position which is consistent with a higher volume state.
Incidence of full stomach on gastric ultrasound assessment | From time of enrollment until the start of surgery, up to 24 hours.
  Incidence of full stomach defined as solid or thick liquids on US or >1.5mL/kg of clear liquid upon gastric ultrasound.
Incidence of regurgitation under anesthesia | From induction of anesthesia until end of surgery (up to 8 hours).
Incidence of change in anesthetic management based on stomach contents | Assessed at enrollment and during gastric ultrasound (within 3 hours of scheduled procedure).
Differences in "high risk GLP-1" vs "low risk GLP-1" | assessed at time of enrollment from the past 30 days until completion of gastric ultrasound
  High Risk includes:
  * Escalation Phase: increase in dose within the past 30 days
  * High Dose
  * Weekly Dosing
  * Presence of severe GI symptoms such as nausea, vomiting, or retching, abdominal bloating, or abdominal pain with GLP-1 administration
  Low dose and high dose are classified as:
  Oral Semaglutide (Rybelsus) Low dose: < 5 mg High dose: > 5 mg
  Tirzepatide (Mounjaro and Zepbound) Low dose: 2.5, 5, and 7.5 mg High dose: 10, 12.5, 15 mg
  SubQ Semaglutide (Ozempic and Wegovy) Low dose: 0.25 and 0.5 mg High dose: 1 and 2 mg
  Dulaglutide (Trulicity) Low dose: 0.75 and 1.5 mg High dose: 3.0 and 4.5 mg
  Liraglutide (Victoza) Low dose: 0.6 mg High dose: 1.2 and 1.8 mg
  Exenatide (Byetta) Low dose: 5 mcg High dose: 10 mcg

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Wolla, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No